CLINICAL TRIAL: NCT01657916
Title: 5-Year Objective and Subjective Results of a Mid-Urethral Sling
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Other Study IDs: R12-01-005
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Stress Urinary Incontinence
Keywords: mid-urethral sling; Align urethral support system; tension free vaginal tape; cough stress test; pelvic exam; PFDI-20; PFIQ; SSQ; Urinary retention; mesh erosion; urodynamics
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 5 year sling implants: Patients who underwent implant of the Align Urethral Support System between June 2007 and December 2008

SUMMARY:
Evaluate 5-year objective and subjective cure rates after implant of the retropubic Align Urethral Support System.

DETAILED DESCRIPTION:
Between June 2007 and December 2008, the investigators performed 155 Align mid-urethral slings in patients who were only receiving this operation. Very few studies have outcomes at 5 years of greater. The aim of this prospective cohort study is to evaluate five-year objective and subjective cure rates. Secondary endpoints will assess failure risk factors and describe any complications of the retropublic Align Urethral Support System five years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* women
* complaint of stress urinary incontinence
* underwent Align urethral support system from June 2007-December 2008

Exclusion Criteria:

* concommitant procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women who suffered from stress urinary incontinence (leakage of urine will laughing/coughing/sneezing/exercising)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Cough stress test | 5 year follow up appt
  Patient will void and their post-void residual amount of urine will be obtained by a catheter. That same catheter will be left in place and used to fill the bladder with 250ml sterile saline. The patient will then be asked to vigorously cough in the upright sitting and standing positions. A positive "cough test" will be defined as any leakage of urine that is visualized during coughing in the sitting or standing position.

SECONDARY OUTCOMES:
Pelvic exam | 5 year follow up appt
  Standardized pelvic exam will be performed to assess healing, palpability, mesh related pain and erosion of the sling.
Stress urinary incontinence related symptoms | 5 year follow up appointment
  Validated stress urinary incontinence related questionnaires were completed prior to surgery by all of these patients, and will be completed 5 years after surgery as well. The specific forms used will be PFDI-20 and incontinence severity index. Question 17 of the pelvic floor distress inventory will be used to assess subjective cure.
Urgency incontinence related symptoms | 5 year follow up appointment
  Patients will be assessed for de novo, stable and improved urgency incontinence using the IIQ-7 subject of PFDI-20 (questions 15, 16, and 18).
Quality of life and self-reported data | 5 year follow up appointment
  Validated questionnaires (Incontinence outcome questionnaire, surgical satisfaction questionaire) will be used to assess patient's surgery satisfaction, subjective self-assessment before and 5 years after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States